CLINICAL TRIAL: NCT03647774
Title: Long Acting Naltrexone for Opioid Addiction: the Importance of Mental, Physical and Societal Factors for Sustained Abstinence and Recovery
Brief Title: Long Acting Naltrexone for Opioid Addiction: Focus on Sustained Abstinence and Recovery
Acronym: NaltRec
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Tanum (Other)
Collaborators: Haukeland University Hospital (Other); Hospital of Southern Norway Trust (Other); The Hospital of Vestfold (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Lars Tanum, Head of Research Unit, R&D dept.in Mental Health, University Hospital, Akershus
Organization: University Hospital, Akershus (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004706-18; 269864 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2018-08-03; First posted 2018-08-27 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Opioid-use Disorder
Keywords: Extended release naltrexone; Opioid dependence; Recovery; Health economics
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Intervention Model Description: A multicenter, open-label treatment study. Extended-release naltrexone hydrochloride injectable suspension (Vivitrol®) (later referred to as XR-NTX) 380 mg/4 weeks One control group enrolled in the national ART program receives "treatment as usual"; flexible dose of daily oral buprenorphine or buprenorphine-naloxone in line with the clinical guidelines in Norway
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Extended release naltrexone (Experimental): Extended release naltrexone 380 mg as an intramuscular injection every 4 weeks.
  Interventions: Drug: Extended release naltrexone
- Treatment As Usual (TAU) (No Intervention): Daily sublingual buprenorphine in flexibel dose according to the patients need and ART guidelines.

INTERVENTIONS:
Drug: Extended release naltrexone — 380mg injectable extended release naltrexone every four weeks
  Other Names: Vivitrol
  Arms: Extended release naltrexone

SUMMARY:
This study is designed as an open-label evaluation of how treatment with XR-NTX may influence the quality and speed of recovery of opioid dependent individuals - in a context of a naturalistic clinical treatment of opioid dependence. The study will assess recovery outcomes and compare these with the clinical effectiveness of XR-NTX (use of illicit substances and safety). Further, the study will assess the recovery outcomes in matched controls receiving treatment with buprenorphine or buprenorphine-naloxone and enrolled in the national OMT program, and compare this with participants receiving XR-NTX.

DETAILED DESCRIPTION:
This is a multicenter, open-label, treatment study of how treatment with extended-release naltrexone hydrochloride injectable suspension (Vivitrol®) (later referred to as XR-NTX) 380 mg/4 weeks will influence or promote the psycho-social recovery and somatic and psychiatric health in opioid dependent individuals. Further the study will investigate the effectiveness and safety of XR-NTX treatment given in a naturalistic setting as an alternative to OMT. The study period is 24 weeks, a subsequent 28 week follow up study and a 1 year post-treatment study. The study is composed of four"Work Packages" (WP). From the same participating sites, a control group of 150 subjects matched on age and gender and currently enrolled in the OMT program receiving daily treatment with either oral buprenorphine or buprenorphine-naloxone will be recruited. Controls will be compared with study participants on psycho-social aspects of recovery and mental and somatic health.

WP1 will use XR-NTX in a clinical naturalistic setting to describe change or improvement in recovery and in illicit drug use for this novel treatment of opioid dependent subjects. A total of n=150 participants will be recruited from five urban hospitals and community health services in Norway to receive treatment with XR-NTX. From the same hospitals and community health services we will also recruit a control group of 150 subjects matched on age and gender already enrolled in the OMT and receiving flexible dose of buprenorphine or buprenorphine-naloxone. The control group will be used for outcomes related to psycho-social recovery and health issues only. There will not be any comparison of use of illicit substances between the XR-NTX and control group. After inclusion in the study and a baseline assessment, the XR-NTX subjects will be followed-up on a monthly basis by the Principal investigator or delegated site personnel. At each visit an injection of XR-NTX will be administered and through an interview, data will be obtained on the use of heroin and other illicit substances, physical and mental health, housing and family situation, income and other social aspects. A urine or saliva sample will be obtained at every visit and screened for opioids and other illicit substances. Fertile women will in addition be screened for pregnancy. All participants will be followed up at 6 and 12 months post-treatment.

The comparison group will be assessed at baseline, after 24 weeks and after 52 weeks only. Study personnel will not administer any medication to subjects in the comparison group.

From XR-NTX participants, a saliva sample will be obtained at baseline (or at a later visit) for genetic analyses to identify possible genetic biomarkers that may predict the outcome of treatment with XR-NTX and possible markers of low catecholaminergic expression (ADHD-spectrum) Community health services from each catchment area that facilitate the recovery process involving community- and specialized health services, will be invited to participate in the study to assess the XR-NTX participants' recovery process every 4 weeks.

Controls will be assessed by the same community health services on their longer term recovery process at week 24 and at week 52.

Assessment of the descriptive elements in the participant's recovery process will be performed using brief structured interviews with the involved health-and social workers. Interviews can be done by telephone or on the net such as teleconference, if feasible.

WP 2 will use qualitative interviews to investigate the subjects' perspective on enablers and barriers to agreeing to and remaining in treatment with, a long-acting opioid receptor antagonist (XR-NTX), including possible emotional reactions and psycho-social implications of treatment. Data will be collected through a) individual semi-structured interviews with approximately 40 of the 150 XR-NTX participants: 20 subjects who stay in treatment for more than 12 weeks and 20 subjects who receive at least one injection XR-NTX but drop out before 12 weeks. In addition, individual interviews and focus group interviews, each with 6-8 close relatives of study subjects will be performed in order to investigate their conceptions regarding the recovery process of their opioid addicted family member; possible changes in familial cohesion and social relationships, and their own need for support and follow-up.

WP 3 is a health-economic study on the cost of XR-NTX treatment in study participants compared to treatment with buprenorphine or buprenorphine-naloxone (OMT) in the controls. Since the cost of medication is only one part of the total health cost of opioid dependence, we will try to estimate the total cost of health- and social services for this group of participants based on national registry data, hospital records and records from GPs and social workers. Registry-based information will be collected based on participants' personal identity number (PIN).

WP4 is designed to increase the knowledge on how opioid receptor antagonism with XR-NTX affects stress, pain and reward responses in patients. WP4 will use specifically measurements of physiological and behavioural responses to stimuli known to be modulated by the brain's opioid system such as social stressors, physical pain and rewards. In addition, data on personality and history of adverse events during childhood that may also be important predictors for adherence to treatment will be collected.

ELIGIBILITY:
Inclusion Criteria:

-.Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

* .Male or female at 18-65 years
* Has a current diagnosis of opioid dependence, based on the criteria of the DSM-V (304.00) as confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* Is voluntarily seeking treatment for opioid dependence
* Completing a stay in a controlled environment with restricted access to substances of abuse with a minimum duration of seven days (waived for OMT controls)
* Is enrolled in the Norwegian national opioid maintenance treatment (OMT) program 'LAR' before discharge from a controlled environment. For subjects who complete & submit their LAR application while in a controlled environment, the investigator may complete enrolment data collection while awaiting response on LAR admission.
* If female and of childbearing potential, must agree to use ahighly effective method of contraception for the duration of the study (waived for OMT controls)
* Capable of understanding and complying with the study procedures

Exclusion Criteria:

* Pregnancy (ie, positive urine and/or serum pregnancy test) and/or currently breastfeeding
* Clinically significant medical condition or observed abnormalities that need medical attention and follow-up (including: severe hepatic (Child-Turcotte-Pugh level C) or renal failure, clinically significant symptoms of progressive Acquired Immunodeficiency Syndrome (AIDS))
* Severe psychiatric disorder (including: current or recurrent affective disorders with suicidal behavior, psychotic disorders) that need medical attention and follow-up
* Use of any excluded medication at screening or anticipated/required use during the study period (including: requiring treatment with opioid medications other than investigational products) (waived for OMT controls)
* Known intolerance and/or hypersensitivity to XR-NTX, carboxymethylcellulose, or polylactide-co-polymers (PLG) or any other components of the diluent (waived for OMT controls).
* Alcoholism defined by the criteria in DSM V
* Serious respiratory debilitation.
* Any finding that in the view of the PI would compromise the subject's ability to fulfill the protocol visit schedule or visit requirements
* Employment by Alkermes or Reckitt-Benckiser (permanent, temporary contract worker, or designee responsible for the conduct of the study) or immediate family of an Alkermes or Reckitt-Benckiser employee.
* Abnormal laboratory assessments. If pathological values, coordinating investigator will decide if the subject is eligible for participation in the study
* Not participating in any other trial that might affect the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Perceived change in recovery | 52 weeks
  Change in recovery assessed by the XR-NTX participant and by their social workers using interview, compared with controls and their social workers.

SECONDARY OUTCOMES:
Use of illicit substances | 52 weeks
  Days of use of illicit opioids and other illicit substances in XR-NTX participants using time-line follow-back every 4th week.
Retention in the study | 52 weeks
  Number of weeks the participants stay in the XR-NTX study (retention)
Craving for heroin | 52 weeks
  Change in craving for heroin in XR-NTX participants using a 100 mm VAS scale, where 0 is no craving and 100 is Maximum craving.
Treatment satisfaction | 52 weeks
  Treatment satisfaction among XR-NTX participants using a 100 mm VAS scale, where 0 is absolutely not satisfactory and 100 is full satisfaction with treatment.
Economic cost analyses | 2 years
  Economic cost analyses across health, community, and criminal justice domains on participants receiving XR-NTX compared to the control group
Change in mental health status | 52 weeks
  Assessment mental health status in participants receiving XR-NTX and controls , measured by the Hopkins'Symptom Check List - 25, a 4-point scale assessing mental distress, 15 depression related items and 10 anxiety related items.
Perceived change in quality of life | 52 weeks
  Change in quality of life assessed by the XR-NTX participant and Controls using the World Health Organization Quality of Life Scale - BREF version, a 24 questions that measure four dimentions of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Tanum, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Loerenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juya F, Klemmetsby Solli K, Sannes AC, Weimand B, Gjerstad J, Tanum L, Mordal J. Genetic Influence on Extended-Release Naltrexone Treatment Outcomes in Patients with Opioid Use Disorder: An Exploratory Study. Brain Sci. 2025 Dec 24;16(1):23. doi: 10.3390/brainsci16010023. PMID 41594744
- [Derived] Mordal J, Juya F, Holtan L, Vederhus JK, Opheim A, Brenna IH, Enger AE, Weimand B, Solli KK, Tanum L. High induction rate onto extended-release naltrexone for people with opioid use disorder: experiences from a Norwegian naturalistic study. Addict Sci Clin Pract. 2025 Jun 16;20(1):50. doi: 10.1186/s13722-025-00576-9. PMID 40524244
- [Derived] Marciuch A, Brenna IH, Weimand B, Solli KK, Tanum L, Rostad BK, Birkeland B. Patients' experiences of continued treatment with extended-release naltrexone: a Norwegian qualitative study. Addict Sci Clin Pract. 2022 Jul 18;17(1):36. doi: 10.1186/s13722-022-00317-2. PMID 35850782